CLINICAL TRIAL: NCT04394793
Title: Low Dose Radiation Therapy for Covid-19 Pneumonia: A Pilot Study
Brief Title: Low Dose Radiation Therapy for Covid-19 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Daya Nand Sharma, Professor, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-AIIMS
Record Dates: First submitted 2020-05-17; First posted 2020-05-19 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Pneumonia
Keywords: Covid-19; pneumonia; low dose radiation therapy
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental)
  Interventions: Radiation: Low dose radiation therapy

INTERVENTIONS:
Radiation: Low dose radiation therapy — Patient will be treated with a dose of 70 cGy in one fraction radiation therapy in addition to standard therapy

SUMMARY:
Radiotherapy in low doses (30 to 100 cGy) was a popular treatment of viral pneumonias until 1940s. Low dose radiation therapy (LDRT) could possibly reduce the inflammation and prevent the cytokine storm thus mitigating the severity of pneumonitis. This is a single arm study designed to assess the feasibility and clinical efficacy of low dose radiation therapy (70 cGy in single fraction) in the patients with COVID-19 pneumonia. A total of 10 eligible patients (as per inclusion criteria) will be recruited and response will be assessed based on the symptomatic improvement or deterioration by using the National Early Warning Score (NEWS). The NEWS score will be recorded on baseline and then on Day 3, Day 7 and Day 14.

DETAILED DESCRIPTION:
There is no specific antiviral treatment recommended for COVID-19, and no vaccine is currently available. The treatment is symptomatic, and oxygen therapy represents the major treatment intervention for patients with severe infection. Mechanical ventilation may be necessary in cases of respiratory failure refractory to oxygen therapy, whereas hemodynamic support is essential for managing septic shock. The death rate ranges from 2-15% in different group of patients.

COVID-19 pandemic is unprecedented in modern history of humankind and it has become imperative to find novel treatments to mitigate the casualties caused by infection. The clinical spectrum of COVID-19 varies from mild symptoms to critical conditions requiring ventilatory support and ICU care. According to Chinese CDC report, 81% patients had mild disease (non-pneumonia and mild pneumonia), 14% had severe disease and 5% had critical disease. Based on severity of symptoms, there are several scoring methods which can predict the outcome of disease. National early warning score (NEWS) is a popular scoring system used for non-ICU patients suffering from acute illness. This score helps in quickly determining the degree of illness and intervention required. It also provides likelihood of death or admission to an ICU. Based on this score any illness can be categorized as mild (Score <4), moderate (Score 5-6 or individual 3) and severe (Score ≥7). According to this scoring system, Covid-19 patients having a score of 5-6 will have probability of 15.7% critical events (HDU/ICU admission or 30-day mortality) and those having score ≥7 will have about 24.1% critical events.

The pathogenesis of COVID-19 pneumonitis appears to involve a cytokine storm with elevated pro- inflammatory cytokines such as IL-6 and TNFα among many others, leading to an onslaught of neutrophils and macrophages, diffuse alveolar damage and respiratory failure. This is where a potential opportunity for low-dose radiation therapy (LDRT) emerges. LDRT is a potential treatment for COVID-19 pneumonia since it has an anti-inflammatory action. Successful management of worsening pneumonia will reduce the development of ARDS and thereby preventing deaths.

Availability of megavoltage beam in modern times has improved our dosimetry in treating deep targets. Radiotherapy which can penetrate lobar and interstitial space can help in preventing both lobar as well as interstitial pneumonia. In the absence of any effective drug and, historical data suggests that low dose of 0.5 to 1 Gy radiotherapy to whole lung can possibly prevent cytokine storm and critical events (ICU admission, mechanical ventilation or death).

The initial use of X-rays to treat patients with pneumonia was reported in 1907. This report offered a new mechanistic insight founded on the dose response, proposing that low doses of X-rays would affect disease resolution. It was observed that not only did the X-ray treatment has lifesaving potential, but it was also effective when other treatments had reached their therapeutic limits as seen in cases of chronic bronchopneumonia, which could be resolved with a single administration of X-rays. Subsequent reports suggested that LDRT was successful in decreasing the mortality rate in untreated patients from about 30% to 5-10%.

Rationale for the Study: It is reasonable to try an LDRT treatment of 30 to 100 cGy to the lungs of a patient with COVID-19 pneumonia as it could reduce the inflammation and relieve the life-threatening symptoms. The recent emerging literature indicates that the efficacy of thoracic LDRT must be investigated as it would present a negligible risk to COVID-19 pneumonia patients, and have the potential to reduce the fatality rates.

Study Design: Interventional, Clinical, Single arm, Pilot study Number of patients: 10 Treatment: Patient will be treated as per COVID-19 standard management protocol of the treating institute along with intervention of Low Dose Radiotherapy (LDRT) 70cGy in single fraction.

Treatment field- Field adequately covering both the lungs. Beam energy : 6MV X-ray photons Number of beams- 2 (1 Anterior and 1 posterior field). Prescription point - Midway of anterior-posterior chest separation. Treatment Workflow: Patients will be maneuvered to lie down on treatment couch in a supine position, with hands above head. Gantry rotated to 90 degree, a lateral chest X ray portal image will be taken, which will guide in measuring dose prescription point. Gantry rotated back to 0 degree; an adequate field size will be opened. Total treatment duration will be about 20-30 minutes.

Response Assessment and statistical analysis: Response will be assessed based on the symptomatic improvement or deterioration by using the NEWS score. The NEWS score will be recorded on baseline and then on Day 3 (D-3), Day 7 (D-7) and Day 14 (D-14). To compare the NEWS score (baseline and post LDRT), student t test (paired) will be used. For statistical significance, p value of 0.1 will be considered significant. Number of patients requiring ICU admission or undergoing death following LDRT will also be recorded to assess critical events.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed cases of Covid-19 (by RT-PCR).
2. Age >18 years.
3. Patients with National Early Warning Score (NEWS) score ≥ 5.
4. Consent

Exclusion Criteria:

1. Patients on mechanical ventilatory support.
2. Hemodynamically unstable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Symptomatic improvement by National Early warning score (NEWS) | Day 3
  NEWS score
Symptomatic improvement by National Early warning score (NEWS) | Day 7
  NEWS score
Symptomatic improvement by National Early warning score (NEWS) | Day 14
  NEWS score
Length of hospital stay | 30 days or date of death whichever is earlier
  Days
Number of ICU admissions or deaths | 30 days
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Daya Nand Sharma, MD, Principal Investigator — AIIMS, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkby C, Mackenzie M. Is low dose radiation therapy a potential treatment for COVID-19 pneumonia? Radiother Oncol. 2020 Jun;147:221. doi: 10.1016/j.radonc.2020.04.004. Epub 2020 Apr 6. No abstract available. PMID 32342871
- [Background] Calabrese EJ, Dhawan G. How radiotherapy was historically used to treat pneumonia: could it be useful today? Yale J Biol Med. 2013 Dec 13;86(4):555-70. PMID 24348219
- [Background] Sbiti-Rohr D, Kutz A, Christ-Crain M, Thomann R, Zimmerli W, Hoess C, Henzen C, Mueller B, Schuetz P; ProHOSP Study Group. The National Early Warning Score (NEWS) for outcome prediction in emergency department patients with community-acquired pneumonia: results from a 6-year prospective cohort study. BMJ Open. 2016 Sep 28;6(9):e011021. doi: 10.1136/bmjopen-2015-011021. PMID 27683509